CLINICAL TRIAL: NCT01551173
Title: A 12-week, Multicenter, Double-blind, Double-dummy, Randomized, Active-controlled, Parallel-group Study to Assess the Efficacy and Safety of Fluvastatin Sodium Extended Release Tablets 80 mg Once Daily Compared to Fluvastatin Sodium Immediate Release Capsules 40 mg Twice Daily (BID) in Chinese Patients With Primary Hypercholesterolemia or Mixed Dyslipidemia at Moderate or High Cardiovascular Risk Who Did Not Achieve Their Lipid Goals When Treated With Fluvastatin Sodium Immediate Release Capsules 40 mg QD
Brief Title: Efficacy and Safety of Fluvastatin Sodium Extended Release Tablets 80 mg Once Daily in Chinese Patients With Primary Hypercholesterolemia or Mixed Dyslipidemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CXUO320BCN01
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Lipid Metabolism Disorders
Keywords: Dyslipidemias; Fluvastatin sodium; Chinese
MeSH Terms: conditions — Lipid Metabolism Disorders; Dyslipidemias | interventions — Fluvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Fluvastatin sodium Extended Release Tablet (Experimental): Oral Fluvastatin sodium Extended Release Tablet 80mg once daily for 12 weeks
  Interventions: Drug: Fluvastatin sodium
- Fluvastatin sodium Immediate Release Capsule (Active Comparator): Oral Fluvastatin sodium Immediate Release Capsule 40mg twice daily for 12 weeks
  Interventions: Drug: Fluvastatin sodium

INTERVENTIONS:
Drug: Fluvastatin sodium — Fluvastatin sodium Extended Release Tablets 80mg

SUMMARY:
This study is to demonstrate therapeutic comparability of Fluvastatin sodium Extended Release Tablets 80 mg QD and Fluvastatin sodium Immediate Release Capsules 40 mg BID in LDL-C lowering from baseline to week 12 (endpoint) in patients with primary hypercholesterolemia or mixed dyslipidemia at moderate or high CV risk who did not achieve their lipid goals when treated with Fluvastatin sodium Immediate Release Capsules 40 mg QD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary hypercholesterolemia or mixed dyslipidemia at moderate or high CV risk according to Chinese Dyslipidemia Guideline (2007).
* Not having achieved lipid treatment goals despite following a cholesterol restrictive diet and/or lipid lowering monotherapy improperly prior to Visit 1 (inclusion in the 6-week open-label study phase).
* Not having achieved lipid treatment goals on a stable dose of Fluvastatin sodium Immediate Release Capsule 40 mg QD during the 6 week open-label study phase (inclusion in the 12-week double-blind study phase).

Exclusion Criteria:

* Patients with known hypersensitivity to fluvastatin or any of the excipients.
* Dyslipidemia secondary to other causes.
* Known muscle disease or history of muscle disease and/or serum CPK levels greater than 2 x upper limit of normal (ULN).
* A history or evidence of Acute Myocardial infarction (AMI), unstable angina (UA) or Coronary artery bypass surgery or Percutaneous Coronary Intervention (PCI) within the previous 8 weeks.
* Active liver disease and/or serum transaminase levels (ALT, AST) greater than 1.5 x ULN.
* Patients on a proper lipid lowering monotherapy (defined as at least 12 weeks continuous monotherapy with a recommended dose and administration in the label) within the previous 3 months prior to visit 1.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Changsha, Hunan, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluvastatin Sodium Extended Release Tablet | Fluvastatin Sodium Immediate Release Capsule
Started | 218 ("Started" indicates randomized) | 218
Full Analysis Set (FAS) | 210 (Patients took at least 1 dose of study drug & had at least 1 post-randomization efficacy parameter) | 214
Completed | 190 | 186
Not Completed | 28 | 32
Not completed — Withdrawal by Subject | 11 | 16
Not completed — Adverse Event | 7 | 6
Not completed — Lost to Follow-up | 5 | 7
Not completed — Other | 5 | 3

BASELINE CHARACTERISTICS:
Population: Randomized Set (RAN)
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluvastatin Sodium Extended Release Tablet | Fluvastatin Sodium Immediate Release Capsule | Total
Number analyzed (Participants) | 218 | 218 | 436
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.8 (8.39) | 60.4 (9.30) | 59.6 (8.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 154 | 296
  Male | 76 | 64 | 140

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in LDL-C From Baseline at Study Endpoint, Week 12 (LOCF)
Description: After the patient has been sitting for at least 5 minutes, a 12 hour fasting blood sample will be withdrawn at baseline and endpoint. An analysis of covariance (ANCOVA) with treatment, center, and indication category as factors and baseline LDL-C as a covariate will be used to analyze percent change from baseline in LDL-C.
Time Frame: Baseline, week 12
Population: FAS: all randomized patients who received at least one dose of double-blind study medication and one post-randomization efficacy parameter measurement. The intent-to-treat principle, patients were analyzed according to the treatment they were assigned to at randomization. Endpoint: final available post-baseline assessment to last scheduled visit
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Fluvastatin Sodium Extended Release Tablet | Fluvastatin Sodium Immediate Release Capsule
Number analyzed (Participants) | 210 | 214
Percent change | -8.692 (1.4229) | -7.887 (1.4258)

2. Secondary Outcome: Change From Baseline at Week 4, Week 8, Week 12, and Endpoint for Lipid Variables Low Density Lipoprotein Cholesterol (LDL-C) , Total Cholesterol (TC), High Density Lipoprotein Cholesterol (HDL-C) , Non HDL-C, Triglycerides (TG)
Description: After the patient has been sitting for at least 5 minutes, a 12 hour fasting blood sample will be withdrawn. An analogous ANCOVA model to that used in the analysis of the primary variable will be used to compare the change in LDL-C, TC, HDL-C, non HDL-C and TG from baseline between treatment groups at Week 4, Week 8, and Week 12
Time Frame: Baseline, week 4, week 8, week 12, Endpoint
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Fluvastatin Sodium Extended Release Tablet | Fluvastatin Sodium Immediate Release Capsule
Number analyzed (Participants) | 210 | 214
mmol/L
  LDL-C week 4 (n=210,214) | -0.447 (0.0427) | -0.438 (0.0426)
  LDL-C week 8 (n=193,194) | -0.418 (0.0460) | -0.408 (0.0465)
  LDL-C week 12 (n=192,189) | -0.353 (0.0475) | -0.377 (0.0485)
  LDL-C Endpoint (n=210,214) | -0.339 (0.0483) | -0.298 (0.0484)
  TC week 4 (n=205,211) | -0.450 (0.0497) | -0.457 (0.0495)
  TC week week 8 (n=193,194) | -0.409 (0.0497) | -0.419 (0.0503)
  TC week 12 (n=192,189) | -0.314 (0.0531) | -0.376 (0.0542)
  TC Endpoint (n=210,214) | -0.294 (0.0548) | -0.290 (0.0549)
  HDL-C week 4 (n=205,211) | -0.004 (0.0118) | 0.002 (0.0118)
  HDL-C week 8 (n=193,194) | 0.012 (0.0128) | 0.016 (0.0130)
  HDL-C week 12 (n=192,189) | 0.034 (0.0129) | 0.010 (0.0132)
  HDL-C Endpoint (n=210,214) | 0.030 (0.0123) | 0.012 (0.0124)
  non HDL-C week 4 (n=205,211) | -0.447 (0.0488) | -0.461 (0.0487)
  non HDL-C week 8 (n=193,194) | -0.422 (0.0484) | -0.438 (0.0490)
  non HDL-C week 12 (192,189) | -0.350 (0.0528) | -0.388 (0.0540)
  non-HDL Endpoint (n=210,214) | -0.325 (0.0550) | -0.305 (0.0551)
  TG week 4(n=205,211) | -0.055 (0.0550) | -0.096 (0.0554)
  TG week 8 (n=193,194) | -0.065 (0.0373) | -0.134 (0.0381)
  TG week 12 (n=192,189) | -0.056 (0.0498) | -0.124 (0.0514)
  TG Endpoint (n=210,214) | -0.031 (0.0559) | -0.088 (0.0566)

3. Secondary Outcome: Proportion of Patients Achieving Their LDL-C Treatment Goals at Week 4, Week 8, Week 12, and Endpoint
Description: LDL-C treatment goal is defined as patients at moderate CV risk with LDL-C levels < 3.37 mmol/L (130 mg/dL) or patients at high CV-risk with LDL-C levels < 2.59 mmol/L (100 mg/dL). The proportion of patients in each treatment group achieving their LDL-C goal during the double-blind period will be compared at Week 4, Week 8, Week 12 and Endpoint using a logistic regression model with treatment and center as factors and baseline LDL-C as a covariate. Odds ratio estimates derived from the logistic regression model and 95%CI will be used to quantify the treatment effect.
Time Frame: Baseline, week 4, week 8, week 12, Endpoint
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | Fluvastatin Sodium Extended Release Tablet | Fluvastatin Sodium Immediate Release Capsule
Number analyzed (Participants) | 210 | 214
Percent of participants
  Moderate cardiovascular risk at week 4 | 50 | 57.1
  Moderate cardiovascular risk at week 8 | 70 | 58.3
  Moderate cardiovascular risk at week 12 | 50 | 54.5
  Moderate cardiovascular risk Endpoint | 50 | 42.9
  high cardiovascular risk at week 4 | 27.2 | 25.9
  high cardiovascular risk at week 8 | 27.9 | 29.1
  high cardiovascular risk at week 12 | 33 | 26.4
  high cardiovascular risk at Endpoint | 31.5 | 24.5

ADVERSE EVENTS:
Groups:
- LescolXL (Fluvastatin Sodium Extended Release Tablet): Oral Fluvastatin sodium Extended Release Tablet 80mg once daily for 12 weeks
- LescolIR (Fluvastatin Sodium Immediate Release Capsule): Oral Fluvastatin sodium Immediate Release Capsule 40mg twice daily for 12 weeks
Arm/Group | LescolXL (Fluvastatin Sodium Extended Release Tablet) | LescolIR (Fluvastatin Sodium Immediate Release Capsule) | Total
Serious Adverse Events (participants affected / at risk) | 4/218 | 2/218 | 6/436
Other Adverse Events (participants affected / at risk) | 18/218 | 14/218 | 32/436
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LescolXL (Fluvastatin Sodium Extended Release Tablet) (N=218) | LescolIR (Fluvastatin Sodium Immediate Release Capsule) (N=218) | Total (N=436)
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 1 | 0 | 1
Drug administration error (Injury, poisoning and procedural complications) | 0 | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0 | 1
Rectal polypectomy (Surgical and medical procedures) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LescolXL (Fluvastatin Sodium Extended Release Tablet) (N=218) | LescolIR (Fluvastatin Sodium Immediate Release Capsule) (N=218) | Total (N=436)
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 3 | 5
Urinary tract infection (Infections and infestations) | 4 | 3 | 7
Blood creatine phosphokinase increased (Investigations) | 4 | 2 | 6
Gamma-glutamyltransferase increased (Investigations) | 2 | 3 | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 3 | 6
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety